CLINICAL TRIAL: NCT03558542
Title: Cardiopulmonary Rehabilitation in Chronic Stroke Patients
Brief Title: Cardiopulmonary Rehabilitation in Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 09.2018.229
Record Dates: First submitted 2018-05-14; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Neurological Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): cardiopulmonary rehabilitation plus neurorehabilitation
  Interventions: Other: cardiopulmonary rehabilitation plus neurorehabilitation

INTERVENTIONS:
Other: cardiopulmonary rehabilitation plus neurorehabilitation — Patients with stroke will undergo an accompanying structured cardiopulmonary rehabilitation program along with a neurorehabilitation program

SUMMARY:
This study is aimed to determine the effects of an accompanying structured cardiopulmonary rehabilitation program along with a neurorehabilitation program on the quality of life, care-giver burden and overall well-being of the patients.

ELIGIBILITY:
Inclusion Criteria:

* A history of ischemic stroke at least 6 months ago

Exclusion Criteria:

* any cardiac or pulmonary problem that renders the patient unavailable for the program
* mental impairment
* not being able to perform exercise testing
* not being able to walk independently

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
VO2max | 2 months
  Maximum oxygen consumption

IPD SHARING:
Plan to Share IPD: No